CLINICAL TRIAL: NCT01689051
Title: Vasodilatory and Metabolic Effects of Glucagon-like Peptide-1 in Periphery Circulation in Patients With and Without Type 2 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Collaborators: Danish Heart Foundation (Other)
Responsible Party: Principal Investigator, Jacob Christian Sivertsen, MD, University Hospital, Gentofte, Copenhagen
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 1-Sivertsen
Record Dates: First submitted 2012-09-17; First posted 2012-09-20 (Estimated); Last update posted 2014-01-31 (Estimated); Status verified 2014-01

CONDITIONS: Type 2 Diabetes; Blod Pressure; Glucagon-like Peptide-1; Human Physiology; Blood Flow
Keywords: Type 2 diabetes; Blod pressure; Glucagon-like peptide-1; Human physiology; Blood flow
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Healthy subjects (Active Comparator)
  Interventions: Other: human glucagon-like peptide 1 (7-36)amide; Other: human glucagon-like peptide 1 (9-36)amide
- Patients with type 2 diabetes (Active Comparator)
  Interventions: Other: human glucagon-like peptide 1 (7-36)amide; Other: human glucagon-like peptide 1 (9-36)amide

INTERVENTIONS:
Other: human glucagon-like peptide 1 (7-36)amide
Other: human glucagon-like peptide 1 (9-36)amide

SUMMARY:
Diabetes and high blood pressure are risk factors for developing heart disease. An increase in the number of diabetes patients is expected. This increases the number of patients with heart disease, and since the vast majority with diabetes die from heart disease, it is extremely important to investigate how these diseases can be prevented and treated.

Studies in animals have shown that intestinal hormone glucagon-like peptide-1 (GLP-1) can expand blood vessels, thus lowering blood pressure, but it is not known whether the effects is found in humans, which we will investigate.

Studies have also shown that GLP-1 lowers blood sugar, but it is unclear whether this is solely due to increased insulin production, weight loss associated with GLP-1 intake or GLP-1 has an effect on the muscles which increases the uptake of sugar. We investigate whether GLP-1 enhances the absorption of sugar in the leg.

The investigators also examines whether these effects are greater in people with diabetes then in healthy.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* T2DM according to WHO's criteria (only T2DM subjects)

Exclusion Criteria:

* Anemia
* T1DM
* Severe liver or renal disease
* Severe heart disease
* Atrial fibrillation

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-03; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Femoral artery blood flow

SECONDARY OUTCOMES:
Leg glucose uptake

CONTACTS AND LOCATIONS:
Overall Officials: Jacob C Sivertsen, MD, Principal Investigator — University Hospital, Gentofte, Copenhagen
Locations (1):
- Gentofte Hospital, Department of Cardiology, Hellerup, Denmark